CLINICAL TRIAL: NCT06758648
Title: Characterizing the Retinal Microvasculature in Patients with Fabry Disease: a Prospective Observational Study
Acronym: VASCinFABRY
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, PD Dr. Christoph Schmaderer, Principal Investigator, Technical University of Munich
Other Study IDs: FD062020
Record Dates: First submitted 2023-04-17; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Fabry Disease; Endothelial Dysfunction; Microvasculature
Keywords: Chronic inflammation; retinal microvasculature; retinal vessel analysis; vasculopathy
MeSH Terms: conditions — Fabry Disease; Vascular Diseases | interventions — Tomography, Optical Coherence; Echocardiography; Pulse Wave Analysis; Blood Pressure Determination; Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are collected from the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Dynamic retinal vessel analysis (DVA) — Dynamic retinal vessel analysis (DVA) is an established, non-invasive technique for evaluating the responsiveness of retinal vessels to flickering light stimuli. This technique allows for the measurement of changes in retinal vessel diameter in response to changes in blood flow, providing insight into the microcirculatory function of the retina. In the case of DVA, patients will asked to focus on a needle, and one arteriole and venule diameter were automatically and continuously recorded. Arteriole and venule segments between 0.5 to 1 mm will be analyzed approximately 2-disc diameters away from the optic nerve in a lower-temporal direction. The baseline recording will be 50 seconds, followed by a flickering phase of 20 seconds and then a recovery period of 80 seconds. Three of these cycles were performed.
  Based on this, we will calculate the percentage of maximum arteriolar (aFID) and venular dilation (vFID) to baseline.
Diagnostic Test: Biochemistry and immune phenotyping — Collection of blood samples from participants for the purpose of performing clinical chemistry analysis. Peripheral blood mononuclear cells (PBMCs) will be isolated from the collected blood samples using standard techniques, such as density gradient centrifugation, and will be analyzed using fluorescence-activated cell sorting (FACS)
Diagnostic Test: Questionnaires (Patient reported outcomes) — This study involves a comprehensive evaluation of life quality, pain, and gastrointestinal (GI) symptoms using a set of established and validated questionnaires. The tools employed include the SF-36 (Short Form-36 Health Survey) to assess overall health-related quality of life across multiple domains, the COMPASS-31 (Composite Autonomic Symptom Score) to evaluate autonomic dysfunction symptoms, and the Brief Pain Inventory (BPI) to measure pain severity and its impact on daily activities. Additionally, the Gastrointestinal Symptom Rating Scale (GSRS) is used to quantify the severity and frequency of GI symptoms, covering dimensions such as reflux, abdominal pain, indigestion, diarrhea, and constipation. Together, these questionnaires provide a multidimensional assessment of the patient's physical, emotional, and symptomatic experiences, allowing for a robust understanding of their health status and quality of life.
Diagnostic Test: Cardio MRI — Cardiovascular magnetic resonance imaging (CMR or cardio MRI) will be utilized in patients with Fabry disease. This imaging technique will enable detailed assessment and monitoring of key cardiac abnormalities, including thickening of the heart walls, left ventricular hypertrophy, and decreased blood flow in the coronary vessels. Additionally, T1 relaxation time measurement will be conducted, offering a non-invasive means to detect myocardial tissue abnormalities such as fibrosis and sphingolipid accumulation, which are hallmarks of Fabry disease. Together, these measures provide a comprehensive evaluation of cardiac structure, function, and tissue characteristics in affected patients.
Diagnostic Test: Optical coherence tomography (OCT) — Optical coherence tomography (OCT) is a non-invasive, high-resolution imaging technique that utilizes low-coherence light to capture cross-sectional images of the ocular fundus. Based on the principle of interferometry, OCT employs low-coherence light, which is scattered by the tissue, to produce detailed, high-resolution images of the retina and its layers. This technology enables precise visualization of the different retinal layers, including the nerve fiber layer, the ganglion cell layer, and the inner and outer plexiform layers. Additionally, OCT can be used to detect and monitor subtle structural changes in the retina, offering critical insights into retinal microarchitecture and potential manifestations of systemic diseases such as Fabry disease.
Diagnostic Test: Echocardiography — Detection of signs of left ventricular hypertrophy, diastolic dysfunction, and valvular disease, which are common cardiac complications associated with Fabry disease, will be a key focus of the assessment. These abnormalities are indicative of the progressive cardiac involvement characteristic of the disease. Left ventricular hypertrophy reflects the thickening of the heart muscle, often caused by sphingolipid accumulation, while diastolic dysfunction highlights impaired relaxation and filling of the left ventricle. Valvular disease, including regurgitation or stenosis, further contributes to the cardiac burden in Fabry disease. Identifying and monitoring these conditions are essential for timely intervention and effective management of cardiac manifestations in affected patients.
Diagnostic Test: 24 hour pulse wave analysis — Pulse wave analysis (PWA) is a non-invasive method used to assess the cardiovascular system. It uses a sensor to measure the pressure waves generated by the heart's contraction and the subsequent blood flow through the peripheral vessels. By analyzing these pressure waves, PWA can provide information about the elasticity of the arterial walls, the blood flow in the peripheral vessels, the blood pressure, and the arterial stiffness.
Diagnostic Test: 24-hour blood pressure measurement — Blood pressure measurement to asses cardiovascular risk.
Diagnostic Test: 1 hour ECG — One hour ECG to asses autonomic dysfunction in patients with Fabry disease.
Diagnostic Test: Ophthalmological consultation — Evaluation and monitoring of ocular manifestations of Fabry disease.
Diagnostic Test: Static retinal vessel analysis (SVA) — Comparable to DVA, SVA is a non-invasive and quick tool to examine the retinal microvasculature. SVA pictures will be analyzed using Vesselmap 2® (IMEDOS Systems GmbH, Jena, Germany). One eye will be examined, and three images will be taken with a focus on the optic disc at an angle of 50°. Roughly one disc diameter away from the optic disc, retinal veins and arterioles segments will be semi-automatically labeled. The Paar-Hubbard formula averages the central retinal arteriolar (CRAE) and central venular (CRVE) equivalents.
  The arteriolar-venular ratio will be calculated as CRAE/CRVE.

SUMMARY:
This study aims to gain a deeper understanding of endothelial dysfunction in patients with Fabry disease through a prospective study of the retinal microvasculature and to identify an objective, non-invasive marker to assess disease severity and cardiovascular risk in patients.

The main questions addressed are: Do dynamic and static retinal vessel analysis parameters differ from those in healthy individuals? Can these parameters predict cardiovascular and/or Fabry-related events during follow-up? Do these parameters change during follow-up in patients with a non-stable disease?

DETAILED DESCRIPTION:
Fabry disease is a rare genetic disorder characterized by the pathological accumulation of glycosphingolipids, specifically globotriaosylceramide (Gb3), within lysosomes in various cells of the body. This accumulation leads to damage in the cardiovascular, cerebrovascular, and renal systems and is characterized by dysfunction of endothelial cells. This dysfunction results in disturbances in the microcirculation and damage to the supplied systems, leading to a significantly increased cardiovascular risk in patients with Fabry disease. Studies have shown that these patients have a higher risk of premature death due to these risk factors compared to the general population.

Early diagnosis and adequate monitoring of enzyme replacement therapy (ERT) are crucial in reducing the risk of cardiovascular events associated with Fabry disease. Currently, LysoGb3 (lysosphingolipid globotriaosylceramide) is considered a biomarker for the diagnosis and monitoring of Fabry disease. Elevated levels of LysoGb3 have been observed in the blood of patients with Fabry disease, and its measurement has been proposed as a diagnostic tool. Additionally, measuring LysoGb3 levels before and after treatment with ERT can be used as a tool to monitor the effectiveness of the therapy in reducing the accumulation of glycosphingolipids in cells and improving symptoms and outcomes in patients with Fabry disease.

However, the performance of LysoGb3 as a predictor of cardiovascular events in patients with Fabry disease is not well understood, and more research is needed to confirm its utility in this regard.

Therefore, there is a need for additional reliable measurements of the microcirculation that can be performed non-invasively and represent a low burden for participants. The use of non-invasive markers of microcirculation can aid in the early diagnosis and monitoring of Fabry disease, which is crucial for the effective use of ERT.

In summary, this study aims to validate new microcirculation markers that can be measured non-invasively in a prospective cohort of patients with Fabry disease and to correlate these markers with established clinical and laboratory parameters. By validating these markers, the study seeks to improve the management of Fabry disease, reduce the burden on participants, and ultimately reduce the incidence of cardiovascular events associated with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Diagnosis of Fabry disease by genetic testing or GB3 activity in leukocytes.
* Signed informed consent form

Exclusion Criteria:

* Active infection or cancer
* Surgery less than 2 weeks prior to inclusion in the study
* Known glaucoma
* Lack of capacity to give consent; lack of informed consent.
* Known epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this study are recruited through our in-house metabolic outpatient clinic (Stoffwechselambulanz), which specializes in the diagnosis, treatment, and long-term management of rare metabolic disorders, including Fabry disease. The clinic serves as a comprehensive care center, offering multidisciplinary services such as genetic counseling, laboratory diagnostics, and individualized treatment planning. Patients are identified and approached during routine follow-ups or initial consultations after confirmation of a Fabry disease diagnosis through genetic testing or measurement of globotriaosylceramide (Gb3) activity in leukocytes. This structured recruitment process ensures the inclusion of well-characterized patients who meet the study's eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Retinal Arteriolar Diameter (CRAE) | From enrollment (T0) to the occurrence of death or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4.
  What will be measured: Central Retinal Arteriolar Equivalent (CRAE) in micrometers (µm).
  Unit of Measure: Micrometers (µm). How it will be reported: Mean CRAE values at baseline for Fabry disease patients compared with age- and sex-matched healthy controls.
Change in Retinal Arteriolar Diameter (CRVE) | From enrollment (T0) to the occurrence of death or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4.
  What will be measured: Central Retinal Arteriolar Equivalent (CRVE) in micrometers (µm).
  Unit of Measure: Micrometers (µm). How it will be reported: Mean CRAE values at baseline for Fabry disease patients compared with age- and sex-matched healthy controls.
Change in arteriolar-venular ration (AVR) | From enrollment (T0) to the occurrence of death or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4.
  What will be measured: AVR as a quotient out of CRAE/CRVE Unit of Measure: no unit How it will be reported: Mean or Median AVR values at baseline for Fabry disease patients compared with age- and sex-matched healthy controls.
Change in Flicker-Induced Venular Dilation (vFID) | From enrollment (T0) to the occurrence of death or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4
  What will be measured: Maximum percentage change in retinal venular diameter during flicker stimulation.
  Unit of Measure: Percentage (%). How it will be reported: Mean vFID percentage change at baseline for Fabry disease patients compared with age- and sex-matched healthy controls.
Change in Flicker-Induced Venular Dilation (aFID) | From enrollment (T0) to the occurrence of death or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4
  What will be measured: Maximum percentage change in retinal arteriolar diameter during flicker stimulation.
  Unit of Measure: Percentage (%). How it will be reported: Mean vFID percentage change at baseline for Fabry disease patients compared with age- and sex-matched healthy controls.
Predictive Value of SVA and DVA Parameters in Fabry Disease Outcomes | From enrollment (T0) to the occurrence of death /FACE or the end of the study, whichever comes first, assessed over an estimated period of up to 4 years. Measurements will be conducted annually, starting at T0, then at 1 year (T1), 2 year (T2), T3 and T4
  What will be measured: The predictive value of Static Retinal Vessel Analysis (SVA) parameters (CRAE, CRVE, AVR) and Dynamic Retinal Vessel Analysis (DVA) parameters (vFID, aFID) in forecasting Fabry disease-associated events (FACE) FACE are measured as preciously described (https://pmc.ncbi.nlm.nih.gov/articles/PMC10359570/) Unit of Measure: Micrometers (µm) for CRAE, CRVE; unitless ratio for AVR; percentage (%) for vFID and aFID.
  Measurement Tools: Retinal vessel analyzers (Static Retinal Vessel Analyzer and Dynamic Retinal Vessel Analyzer, IMEDOS Systems, Jena, Germany), echocardiography, clinical laboratory markers (e.g., LysoGb3), and DS3 scoring system. FACE.
  How it will be reported Hazard Ratios (HR): Derived from Cox proportional hazard models Odds Ratios (OR): For binary outcomes Multivariable Regression Models
  Receiver Operating Characteristic (ROC) Analysis:
  Correlation Coefficients: (e.g., Pearson or Spearman)

SECONDARY OUTCOMES:
Correlation Between Retinal Vessel Parameters and Symptom Severity (DS3) | Measurement at enrollment (T0)
  What will be measured: Correlation of static retinal vessel analysis parameters (CRAE, CRVE, AVR) and dynamic parameters (vFID, aFID) with the Fabry disease severity score (DS3, Giannini et al. 2009).
  Unit of Measure: Micrometers (µm) for CRAE, CRVE, AVR; percentage (%) for vFID and aFID; unitless for DS3 score (range 0-32).
  Measurement Tools: Dynamic Retinal Vessel Analyzer (IMEDOS Systems, Jena, Germany), Static Retinal Vessel Analyzer (IMEDOS Systems, Jena, Germany), and the DS3 scoring system.
  How it will be reported: Statistical correlation coefficients (e.g., Spearman or Pearson).
Patients with Fabry disease and impaired retinal microcirculation Elevated Markers of Endothelial Dysfunction and Chronic Inflammation in Patients With Impaired Retinal Microcirculation | Measurement at enrollment (T0)
  What will be measured: Concentration of markers of endothelial dysfunction (sICAM, sVCAM, Thrombomodulin, P-Selectin, E-Selectin, ADMA, SADMA, Endothelin-1) and chronic inflammation (IFN-β, IFN-λ1, TNF-α).
  Unit of Measure: Nanograms per milliliter (ng/mL) for most markers; other units (e.g., µmol/L for ADMA) as specified.
  Measurement Tools: ELISA, flow cytometry (e.g., FACS analysis for PBMCs). How it will be reported: Mean concentrations or median with interquartile range (IQR).
Correlation Between Retinal Microcirculation Markers and Cardiac Damage | Measurement at enrollment (T0)
  What will be measured: Static retinal vessel analysis parameters (CRAE, CRVE, AVR) and dynamic parameters (vFID, aFID) correlated with cardiac measurements ( thickness of interventricular septum, posterior wall thickness, left ventricular end diastolic diameter) and incidence of cardiovascular events (e.g., heart failure, arrhythmia).
  Unit of Measure: Micrometers (µm) for retinal vessel parameters; millimeters (mm) for cardiac measurements.
  Measurement Tools: Retinal vessel analyzers (IMEDOS Systems, Jena, Germany) and echocardiography.
  How it will be reported: Statistical correlation coefficients (e.g., Spearman or Pearson).
Correlation Between Genetic Phenotypes and Retinal Vessel Parameters | Measurement at enrollment (T0)
  What will be measured: Static retinal vessel analysis parameters (CRAE, CRVE, AVR) and dynamic parameters (vFID, aFID) correlated with genetic classifications (classical, non-classical Fabry disease) and pathogenicity of GLA gene variants.
  Unit of Measure: Micrometers (µm) for retinal vessel parameters; categorical classifications for genetic phenotypes (classical, non-classical).
  Measurement Tools: Retinal vessel analyzers (IMEDOS Systems, Jena, Germany) and genetic analysis using ACMG guidelines.
  How it will be reported: Mean retinal parameters for each genetic phenotype group; statistical correlations.
Polymorphisms in the Human Endothelial Nitric Oxide Synthase Gene (eNOS) | Measurement at enrollment (T0)
  What will be measured: Frequency and type of gene polymorphisms in the human endothelial nitric oxide synthase (eNOS) gene.
  Unit of Measure: Proportion of participants (%) with specific polymorphisms. Measurement Tools: Polymerase chain reaction (PCR) and restriction fragment length polymorphism (RFLP) analysis.
  How it will be reported: Percentage of participants with each polymorphism type.
Comparison of Vessel Density in OCT-A Between Fabry Patients and Healthy Cohort | Measurement at enrollment (T0)
  What will be measured: Vessel density in the retina using optical coherence tomography angiography (OCT-A).
  Unit of Measure: Percentage (%) of vessel density. Measurement Tools: Optical coherence tomography angiography (OCT-A). How it will be reported: Mean vessel density values for Fabry patients versus healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Günthner, PD Dr., Principal Investigator — Abteilung für Nephrologie; Timon Kuchler, Principal Investigator — Abteilung für Nephrologie; Matthias Braunisch, Pd Dr., Principal Investigator — Abteilung für Nephrologie; Claudia Regenbogen, Study Chair — Abteilung für Nephrologie; Christoph Schmaderer, Study Director — Abteilung für Nephrologie
Locations (1):
- Department of nephrology, Klinikum rechts der Isar, München, Bavaria, Germany

REFERENCES:
- [Background] Giannini EH, Mehta AB, Hilz MJ, Beck M, Bichet DG, Brady RO, West M, Germain DP, Wanner C, Waldek S, Clarke JT, Mengel E, Strotmann JM, Warnock DG, Linhart A. A validated disease severity scoring system for Fabry disease. Mol Genet Metab. 2010 Mar;99(3):283-90. doi: 10.1016/j.ymgme.2009.10.178. Epub 2009 Oct 30. PMID 19951842
- [Background] Hughes DA, Bichet DG, Giugliani R, Hopkin RJ, Krusinska E, Nicholls K, Olivotto I, Feldt-Rasmussen U, Sakai N, Skuban N, Sunder-Plassmann G, Torra R, Wilcox WR. Long-term multisystemic efficacy of migalastat on Fabry-associated clinical events, including renal, cardiac and cerebrovascular outcomes. J Med Genet. 2023 Jul;60(7):722-731. doi: 10.1136/jmg-2022-108669. Epub 2022 Dec 21. PMID 36543533
- [Derived] Wallraven T, Regenbogen C, Gunthner R, Ribeiro A, Carbajo-Lozoya J, Hannane N, Wunderle M, Assaf A, Lech M, Hanssen H, Streese L, Hughes D, Haller B, Kotliar K, Heemann U, Schmaderer C. Endothelial dysfunction in Fabry disease: retinal biomarkers link cardiac GLA gene variants with chronic inflammation. NPJ Genom Med. 2026 Jan 16. doi: 10.1038/s41525-025-00540-1. Online ahead of print. PMID 41545379